CLINICAL TRIAL: NCT05542017
Title: Long-term Outcome Following Concomitant Surgical Ablation for Atrial Fibrillation at University Hospital Basel: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Elodie Hersperger, Principal Investigator, University Hospital, Basel, Switzerland
Other Study IDs: 2018-00206
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation; Maze Procedure
Keywords: Surgical Ablation; Cardiac Surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgical Ablation for Atrial Fibrillation — Surgical ablation in combination with other cardiac procedures through a median sternotomy or thoracotomy. Main procedures were valve surgery (i.e. repair, replacement) and/or coronary artery bypass grafting (CABG). Surgical ablation procedures for atrial fibrillation were divided into three different groups according to Heart Rhythm Society (HRS) expert consensus 2017: (1) Pulmonary vein isolation alone; (2) Pulmonary vein isolation combined with left atrial lesion sets; (3) and biatrial procedure.

SUMMARY:
This retrospective single-centre study aims to examine the success rate of concomitant surgical ablation in patients with atrial fibrillation (AF) with an up to eight years follow-up period. Moreover, the focus of this study was to identify variables which predict freedom from AF, such as the type of AF, lesion set performed, energy source used and the patient's characteristics.

ELIGIBILITY:
Inclusion Criteria:

* concomitant surgical ablation for atrial fibrillation
* performed between January 2011 and January 2017 at University Hospital Basel

Exclusion Criteria:

* stand-alone procedure
* surgical ablation for atrial flutter

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent concomitant surgical ablation for atrial fibrillation between January 2011 and January 2017 at the University Hospital of Basel. The study population consisted of patients with paroxysmal, persistent, and long-standing persistent AF as defined by the 2020 ESC-Guidelines. Surgical ablation was performed concomitant to cardiac surgery addressing valvular or ischemic heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Freedom from AF one year after surgical ablation | 12 months
  one-year success

SECONDARY OUTCOMES:
Freedom from atrial fibrillation (AF) and atrial flutter (AFL) after removal from antiarrhythmic drug therapy | from surgical ablation until 10th October 2019
Need of additional arrhythmia interventions | from surgical ablation until 10th October 2019
  repeat ablation procedures, electrical cardioversion, pacemaker implantation or implantable cardioverter-defibrillator (ICD) implantation
Use of oral anticoagulation | from surgical ablation until 10th October 2019
Perioperative morbidity | from surgical ablation until 10th October 2019
Mortality | from surgical ablation until 10th October 2019
Evolution of left atrial size | from surgical ablation until 10th October 2019

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation: Executive summary. Europace. 2018 Jan 1;20(1):157-208. doi: 10.1093/europace/eux275. No abstract available. PMID 29016841